CLINICAL TRIAL: NCT06533722
Title: A Phase II Study of the Efficacy and Safety of Adaptive Therapy for Metastatic Refractory Breast Cancer
Brief Title: Adaptive Therapy for Post-Second-Line Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-049
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HER2-negative Metastatic Breast Cancer
MeSH Terms: interventions — Gemcitabine; Vinorelbine; eribulin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Gemcitabine Gemcitabine 1000 mg/m^2 IV on days 1 and 8, cycled every 33 days Vinorelbine 25 mg/m^2 IV on days 1 and 8, cycled every 33 days Eribulin 1.4 mg/m^2 IV on days 1 and 8, cycled every 33 days
  Interventions: Drug: Gemcitabine, Vinorelbine, or Eribulin

INTERVENTIONS:
Drug: Gemcitabine, Vinorelbine, or Eribulin — Gemcitabine Gemcitabine 1000 mg/m^2 IV on days 1 and 8, cycled every 33 days Vinorelbine 25 mg/m^2 IV on days 1 and 8, cycled every 33 days Eribulin 1.4 mg/m^2 IV on days 1 and 8, cycled every 33 days
  Other Names: chemotherapy

SUMMARY:
The primary objective of this study is to explore the efficacy and safety of adaptive therapy in the treatment of post-second-line metastatic breast cancer.

DETAILED DESCRIPTION:
This is a phase II, prospective, single arm clinical trial. The objective of the study is to evaluate the efficacy and safety of adaptive therapy in the treatment of post-second-line advanced breast cancer. The therapy regimen primarily including Gemcitabine, Vinorelbine, or Eribulin, will be selected by the investigator based on current guidelines, available treatments, and an assessment of the patient's clinical status, preferences, and financial situation. This study plans to recruit 10 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Understands and voluntarily signs the informed consent form.
* Minimum life expectancy 16 weeks.
* Histologically or cytologically confirmed advanced invasive breast cancer.
* Histological type: human epidermal growth factor receptor 2 (HER2) negative.
* Prior failure of at least first-line treatment for metastatic disease.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Adequate organ function including bone marrow, renal function, hepatic function, and cardiac reserve.
* Premenopausal women must use medically acceptable contraception during the study.
* Compliance with the study protocol.

Exclusion Criteria:

* Pregnant or breast feeding.
* Uncontrolled medical problems.
* Evidence of active acute or chronic infection.
* Hepatic, renal, cardiac, or bone marrow dysfunction.
* Concurrent malignancy or history of other malignancy within the last five years.
* Patients were unable or unwilling to comply with program requirements.
* Concurrent use of any other anti-cancer therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months
  The interval time from the date of initiation treatment after recruit to the date of the first documented disease progression or death due to any cause.

SECONDARY OUTCOMES:
Occurrence and severity of adverse events (AEs) | 12 months
  Occurrence and severity of AEs by NCI-CTCAE v5. Changes in laboratory parameters (hematology and serum chemistry), vital signs and ECG parameters. Grade 3 or 4 abnormalities in serum chemistry laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No